CLINICAL TRIAL: NCT05094193
Title: Trocar-site Infiltration With Ropivacaine Versus Tranversus Abdominis Plane Block Following Laparoscopic Cholecystectomy: a Double-blinded, Randomized-controlled Trial
Brief Title: Trocar-site Infiltration Versus TAP-block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Daghmouri Mohamed Aziz, Principal investigator, Tunis University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HTHEC-2021-29
Record Dates: First submitted 2021-10-03; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Acute pain management; Ropivacaine; Trocar-site infiltration; TAP-block; Laparoscopic cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trocar-site infiltration (Experimental): Trocar-site infiltration with 20 mL of ropivacaine 0.375% (6 mL in 10 mm trocar site and 4 mL in 5 mm trocar site) associated with bilateral TAP block with 20 mL of normal saline in each side
  Interventions: Procedure: Trocar-site infiltration; Procedure: TAP block placebo
- TAP block (Active Comparator): Trocar-site infiltration with 20 mL of normal saline associated with bilateral TAP block with 20 mL of ropivacaine 0.375% in each side
  Interventions: Procedure: TAP block; Procedure: Trocar site infiltration placebo

INTERVENTIONS:
Procedure: Trocar-site infiltration — 20 mL of ropivacaine 0.375% (6 mL in 10 mm trocar site and 4 mL in 6 mm trocar site)
  Arms: Trocar-site infiltration
Procedure: TAP block — bilateral ultrasound-guided TAP block with 20 mL of ropivacaine 0.375% in each side
  Arms: TAP block
Procedure: Trocar site infiltration placebo — 20 mL of normal saline
  Arms: TAP block
Procedure: TAP block placebo — bilateral ultrasound-guided TAP block with 20 mL of normal saline in each side
  Arms: Trocar-site infiltration

SUMMARY:
For symptomatic gall bladder disorders (cholelithiasis and cholecystitis), laparoscopic cholecystectomy (LC) has been considered as the gold standard treatment. However, these minimally invasive technique is associated with acute moderate pain during the 24 hours postoperative, which is routinely managed using opioids. The transversus abdominis plane (TAP) block has been used as part of a multimodal analgesia strategy. Besides, Wang et al found that TAP block is more effective than a conventional pain control, but not significatively different from another local incisional pain control that is port site infiltration.So, the aim of this study, is to compare the analgesic efficacy and safety of trocar-site infiltration with ropivacaine with ultrasound-guided TAP block following laparoscopic cholecystectomy when used as part of multimodal analgesia.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* Scheduled for laparoscopic cholecystectomy
* ASA grade I, II and III

Exclusion Criteria:

* Bile duct exploration, insertion of a T-drain or patients with acute cholecystitis
* Conversion to open cholecystectomy or if the surgery exceeded 200 minutes
* Severe systemic disease
* Patients on analgesics for any reason
* History of allergy to local anesthetics
* An ongoing pregnancy
* Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain | up to 24 hours
  Visual analog scale (VAS) 0: "no pain" to 10: "severe pain" at rest and cough
Total opioid consumption | Day 1

SECONDARY OUTCOMES:
Length of hospital stay | up to 1 week
postoperative nausea and vomiting | Day 1
Patient satisfaction and quality of recovery | Day 1
  QoR-40 questionnaire
Incidence of shoulder pain | Day 1
Postoperative complication | up to 1 week
  Ileus, wound infection, wound abscess

CONTACTS AND LOCATIONS:
Overall Officials: BEN FADHEL Kamel, M.D, Study Director — Habib Thameur Hospital of Tunis, Department of Anesthesia
Locations (1):
- Habib Thameur Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided